CLINICAL TRIAL: NCT00670228
Title: A Multi-center, Phase 3b, Stratified, Randomized, Open-label Clinical Trial to Evaluate the Efficacy of Intensive Apidra®/Lantus® Therapy vs Sliding Scale Insulin on Infarct Size in Hyperglycemic Subjects With Anterior STEMI (ST Elevation Myocardial Infarction) Undergoing PCI (Percutaneous Coronary Intervention)
Brief Title: Effect of Lantus and Apidra in Patients With Acute ST Elevation Myocardial Infarction
Acronym: INTENSIVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to Negative feasibility assessment of recruiting the planned number of subjects within the study timelines
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_01687
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-01

CONDITIONS: AMI
MeSH Terms: interventions — Insulin Glargine; insulin glulisine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Insulin Therapy (IIT) (Active Comparator): In IIT arm, subjects received intravenous (IV) insulin glulisine and subcutaneous (sc) insulin glargine to maintain a Blood Glucose (BG) concentration between 90-130 mg/dL.
  Interventions: Drug: Insulin Glargine (LANTUS); Drug: Insulin Glulisine (Apidra)
- Standard Glycemic Care (SGC) (Active Comparator): In SGC arm subjects assigned to "standard of care" received subcutaneous regular insulin per sliding scale.
  Interventions: Drug: Standard Therapy

INTERVENTIONS:
Drug: Insulin Glargine (LANTUS) — Subcutaneous insulin glargine was initiated 90 prior to the insulin glulisine infusion discontinuation (i.e. 48 hours after randomization) and titrated as per physician preference to maintain the plasma glucose between 90-130 mg/dL
  Arms: Intensive Insulin Therapy (IIT)
Drug: Insulin Glulisine (Apidra) — Prior PCI, subjects received a single IV bolus of insulin glulisine. The dose was 0.025 U/kg based upon patient reported weight.
  Then IV insulin glulisine infusion was started within one hour of the IV insulin glulisine bolus and administered at a minimum rate of 2 U/h for 48 hours. The infusion was titrated in order to achieve and maintain the plasma glucose between 90 and 130 mg/dL.
  Arms: Intensive Insulin Therapy (IIT)
Drug: Standard Therapy — Standard insulin therapy titrated to blood sugar control
  Other Names: multiple insulins per hospital protocol
  Arms: Standard Glycemic Care (SGC)

SUMMARY:
Primary objective:

To demonstrate that in hyperglycemic subjects with anterior STEMI (ST Elevation Myocardial Infarction) undergoing Percutaneous Coronary Intervention (PCI), tight glycemic control using insulin glulisine and insulin glargine, i.e. Intensive Insulin Therapy (IIT), results in reducing infarct size at day 60 versus (vs) Standard Glycemic Care (SGC).

Secondary objectives:

To demonstrate that tight glycemic control using insulin glulisine and insulin glargine reduces markers of inflammation and improves Left Ventricular (LV) function and Cardio-Vascular (CV) outcomes from baseline values, in hyperglycemic subjects with STEMI undergoing Percutaneous Coronary Intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Men or women = or > 35 years of age presenting to the hospital with hyperglycemia (plasma glucose >140 mg/dL) and Primary Anterior wall ST-Elevation Myocardial Infarction (AW STEMI)
* No history of illicit drug abuse in past year
* A minimum of 30 minutes but < or = 6 hours of continuous pain/symptoms immediately prior to presentation
* Subjects who will undergo primary percutaneous coronary intervention (PCI)
* At least 2 contiguous precordial leads demonstrating at least 2 mm of ST-segment elevation consistent with anterior wall MI
* Signed informed consent and HIPAA documentation (US only) prior to participation in the study
* Subjects ability and willingness to adhere to and be compliant with study protocol

Exclusion Criteria:

* A prior history of Myocardial Infarction (MI)
* Subjects who have received any thrombolytic therapy during the current hospital admission
* Severe Heart Failure or cardiogenic shock (Killip class 3 or 4) by history or present at the time of screening
* Subjects with a plasma glucose >400 mg/dL or diabetic ketoacidosis (DKA)
* History of Type 1 diabetes
* Active bleeding
* Active malignancy, chronic or other medical conditions likely to result in death over the next one year
* Recent hypotension requiring inotropic support in the past 30 days
* Participation in another clinical research study in the past 30 days
* Pregnant or lactating women (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method)
* Unwilling to give informed consent
* Subjects directly involved in the conduct of the study
* Known hypersensitivity to insulin glargine or glulisine
* Contraindication to MRI: a)Intracranial aneurysm clips (Unless the investigator is certain that it is made of non-ferromagnetic material such as titanium)b)Intra-orbital metal fragments c)Any electrically, magnetically or mechanically activated implants (including cardiac pacemakers, biostimulators, neurostimulators, cochlear implants, and hearing aids) d)Warning about Gadolinium-based contrast agents (GBCAs) Exposure to GBCAs increases the risk for nephrogenic systemic fibrosis (NSF). Therefore the following subjects should be excluded from the trial based on a history and/or laboratory tests:

  * acute or chronic severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2), as calculated by the MDRD (Modification of diet in Renal Disease) equation, or
  * acute renal insufficiency of any severity
* Subjects with blood pressure > or = to 200/110 mmHg at time of randomization
* Subjects with a high degree of non-transient AV (Atrio-Ventricular) block

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Operations, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter study: 60 out of the 90 centers planned were initiated. Only 17 centers randomized patients (i.e. 7 sites in the United States, 5 sites in Argentina, 3 sites in Brazil and 2 sites in Mexico).
Pre-assignment Details: Although 34 patients signed the informed consent form for study inclusion, one patient did not sign the Health Insurance Portability and Accountability Act (HIPAA) form, electing to keep his/her medical information private, and was therefore not randomized.
Period: Overall Study
Arm/Group | Intensive Insulin Therapy (IIT) | Standard Glycemic Care (SGC)
Started | 18 | 15
Completed | 13 | 12
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Death or MACE | 0 | 1
Not completed — Not treated | 2 | 2
Not completed — Not meeting the selection criteria | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Insulin Therapy (IIT) | Standard Glycemic Care (SGC) | Total
Number analyzed (Participants) | 18 | 15 | 33
Age Continuous [Mean (Standard Deviation); unit: years] | 61.11 (10.95) | 62.80 (11.12) | 61.88 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 12 | 13 | 25
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — BMI = body weight in kilograms/height in meters squared
  Kg/m^2 | 26.95 (3.34) | 28.49 (3.92) | 27.65 (3.64)
Diabetes diagnosis at study entry [Number; unit: participants]
  Yes | 6 | 7 | 13
  No | 12 | 8 | 20
Duration of Diabetes at study entry [Mean (Standard Deviation); unit: Years] — One data is missing for the Standard Glycemic Care (SGC) arm (n=14 subjects).
  Years | 9.50 (9.20) | 7.50 (6.80) | 8.50 (7.79)
Mean time to Percutaneous Coronary Intervention (PCI) [Mean (Standard Deviation); unit: minutes] | 110.00 (112.69) | 101.54 (51.47) | 106.07 (88.21)
Myocardial Infarction (MI) duration greater than 3 hours [Number; unit: participants]
  No | 13 | 9 | 22
  Yes | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Infarct Size Absolute Change From Baseline at Day 60
Description: Infarct size is measured by cardiac Magnetic Resonance Imaging (MRI) as the percentage of Left Ventricular (LV) mass.
Time Frame: From baseline at Day 60
Population: Analysis was performed on the Modified Intention To Treat (MITT) population which includes all randomized subjects who took at least one dose of the study medication, undergone PCI procedure at hospital admission, and had a valid post-PCI infarct size.
Measure: Mean (Standard Deviation); unit: percentage of LV mass change
Arm/Group | Intensive Insulin Therapy (IIT) | Standard Glycemic Care (SGC)
Number analyzed (Participants) | 11 | 12
percentage of LV mass change | -7.84 (9.19) | -15.72 (22.41)

2. Secondary Outcome: Left Ventricular (LV) Function Evaluated by Cardiac Magnetic Resonance Imaging (MRI)
Description: Due to study early termination and the limited number of randomized subjects, descriptive statistics for the Day 3 Ejection Fraction were selected for presentation instead of for Day 60 as initially planned.
Time Frame: At Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Ejection Fraction
Arm/Group | Intensive Insulin Therapy (IIT) | Standard Glycemic Care (SGC)
Number analyzed (Participants) | 11 | 12
percentage of Ejection Fraction | 43.08 (11.34) | 43.43 (6.87)

3. Secondary Outcome: Occurrence of the Major Adverse Cardiovascular Events (MACE)
Description: MACE:
  Cardiac death, New onset or worsening congestive heart failure (>24 h post-admission) event evaluating using New York Heart Association (NYHA) Class II or greater Non-fatal Myocardial Infarction, Severe arrhythmia, Stroke/TIA (Transient Ischemic Attack), Cardiogenic shock, Catheterization/revascularization, Unstable angina leading to hospitalisation
Time Frame: At Day 60
Population: Analysis was performed on the safety population which includes all subjects who received any study treatment. All subjects in this population were analyzed according to the actual treatment they received.
Measure: Number; unit: events
Arm/Group | Intensive Insulin Therapy (IIT) | Standard Glycemic Care (SGC)
Number analyzed (Participants) | 16 | 13
events
  Severe arrhythmia | 7 | 2
  Shock | 0 | 1
  Revascularization | 1 | 0
  New onset or worsening of congestive heart failure | 1 | 0
  Myocardial Infarction (MI) | 1 | 0
  Death | 1 | 1

4. Secondary Outcome: Biomarkers of Inflammation Measurement: CRP (C-Reactive Protein)
Time Frame: At Day 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Intensive Insulin Therapy (IIT) | Standard Glycemic Care (SGC)
Number analyzed (Participants) | 11 | 12
mg/L | 2.52 (2.10) | 2.96 (4.07)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the first to the last drug intake + 1 week after the administration of the last intake i.e. end of the study.
Arm/Group | Intensive Insulin Therapy (IIT) | Standard Glycemic Care (SGC)
Serious Adverse Events (participants affected / at risk) | 6/16 | 3/13
Other Adverse Events (participants affected / at risk) | 10/16 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Insulin Therapy (IIT) (N=16) | Standard Glycemic Care (SGC) (N=13)
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 1 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 2
Bronchopneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Insulin Therapy (IIT) (N=16) | Standard Glycemic Care (SGC) (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 2
Ventricular Fibrillation (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 1 | 0
Injection Site Phlebitis (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Sudden Cardiac Death (General disorders) | 0 | 1
Venipuncture Site Swelling (General disorders) | 1 | 0
Vessel Puncture Site Haematoma (General disorders) | 2 | 1
Vessel Site Puncture Haemorrhage (General disorders) | 1 | 0
Vessel Puncture Site Pain (General disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Blood Magnesium Decreased (Investigations) | 1 | 0
Transaminases Increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Petechia (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 4 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Only descriptive statistics were presented for primary and key secondary efficacy endpoints. The analysis focused on a review of safety Adverse Events (AEs) data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.